CLINICAL TRIAL: NCT05373550
Title: Effectiveness of a Nursing Educational Intervention on Quality of Life, Sexual Function, and Self-esteem in Hysterectomized Women: a Mixed-method Approach
Brief Title: Effectiveness of a Nursing Intervention on Quality of Life, Sexual Function, and Self-esteem in Hysterectomized Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Concepcion (Other)
Collaborators: Universidad Central del Ecuador (Other)
Responsible Party: Principal Investigator, Alide Salazar Molina, Research director, Universidad de Concepcion
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEBB 717_2020
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Prevention of Complications Due to Hysterectomy
Keywords: Quality of Life; Sexuality; Self Concept; Hysterectomy
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Intervention Model Description: The design will be a sequential exploratory mixed design, which consists of an initial phase of qualitative data collection and analysis and a final phase where quantitative data are collected and analyzed. This mixed mixture allows for clear stages to be determined, with the data from one stage needing to be thoroughly analyzed before the other stage provides details about the intervention study model.
Masking Description: As blinding is a necessary condition in this type of study, the knowledge of the surveyors in the collection of the data, about the experimental group and comparison group will be safeguarded, for which the list of the participating women will be delivered in sealed envelopes and they will only know as group A and group B, both at the beginning and at the end of the study in the pre-test and post-test, with the aim of preventing certain biases in some of the stages of the study, reducing the possibility that the variables of results and their measurement are influenced by lack of blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison group: usual care (No Intervention): It is made up of women between 35 and 65 years old who are on the waiting list for surgical treatment (hysterectomy) of the gynecology service of the HGOLEA and receive routine care.
- Experimentation group: nursing education intervention with technological support. (Experimental): It is made up of women between 35 and 65 years of age who are on the waiting list for surgical treatment (hysterectomy) in the gynecology service of the HGOIA. Women seen at this facility receive care similar to that previously described for the HGOLEA. This group will additionally receive the educational intervention of face-to-face nursing with technological support.
  Interventions: Behavioral: Effectiveness of a nursing educational intervention on quality of life, sexual function, and self-esteem in hysterectomized women: a mixed method approach.

INTERVENTIONS:
Behavioral: Effectiveness of a nursing educational intervention on quality of life, sexual function, and self-esteem in hysterectomized women: a mixed method approach. — Effectiveness of a nursing educational intervention supported by a technological tool (Libre mujer), on quality of life, sexual function and self-esteem in hysterectomized women: a mixed method approach.
  Arms: Experimentation group: nursing education intervention with technological support.

SUMMARY:
Surgical hysterectomy is second only to cesarean section as a surgical procedure in women, causing an impact on sexual function, quality of life, and self-esteem, therefore it is necessary to incorporate a comprehensive care in search of women's welfare.

Objectives: To know the meaning of education in the perioperative period, in women submitted to hysterectomy for a benign cause.

To determine the efficacy of a nursing educational intervention based on self-care in the improvement of sexual function, health-related quality of life, and self-esteem in women undergoing hysterectomy for benign causes.

Subjects and methods: A sequential exploratory mixed-method study. For the qualitative phase, individual interviews will be conducted with women (35 to 65 years old) with the indication of hysterectomy for benign pathology attending the gynecology office, who will be contacted and invited to participate. The interviews will be analyzed using the content analysis technique. The quantitative phase will correspond to a quasi-experimental study design with a non-equivalent control group in women with indications for hysterectomy between 35 and 65 years old in two Obstetric Gynecological Hospitals in Quito. At least 26 women on the waiting list for hysterectomy for the experimental group and 26 for the comparison group will be included.

Instruments: Bio-sociodemographic questionnaire, Female Sexual Function Index, SF-36, and Rosenberg Scale. The two groups will receive traditional care and the experimental group will additionally receive face-to-face nursing educational intervention with technological support.

Ethical requirements will be considered. Expected results: After the nursing education intervention with technological support, women in the experimental group will improve their sexual function, health-related quality of life, and self-esteem concerning the comparison group

DETAILED DESCRIPTION:
TITLE: Effectiveness of a nursing educational intervention on quality of life, sexual function and self-esteem in hysterectomized women: a mixed-method approach.

1.1 PRESENTATION AND RATIONALE OF THE PROBLEM The 20th century has been decisive for the development in different areas of medicine, the great advances achieved have allowed to increase life expectancy at birth and to modify the population pyramids in many countries of the world, reaching in Ecuador 79.30 years in women and 73.33 in men, which has determined that more and more women spend at least a third of their lives after menopause.

However, it is worth mentioning that the physiological transition of menopause can be altered by a surgical procedure to resolve common and more prevalent benign neoplasms such as fibroids, abnormal uterine bleeding, pelvic pressure, among others, inducing surgical or induced menopause in some cases, defined by the Council of Affiliated Menopause Societies (CAMS), of the International Menopause Society, as the definitive cessation of menstruation due to irreversible gonadal damage induced by surgical excision.

Hysterectomy is the most performed major gynecological procedure in the world, becoming a subject of controversy from its beginnings to the present time, therefore, hysterectomy is the last decision in the treatment of gynecological problems and leads the woman to a long period of symptoms for the final decision.

Although most hysterectomies are performed to improve the woman's quality of life, their impact has not been adequately measured and can be markedly heterogeneous, with reports of beneficial, negative, and neutral effects.

Thus, it has been described that the radicality of surgical or induced menopause has an impact on the quality of life, altering femininity, causing physical, psychological, social, and sexual well-being alterations, accounting for a subjectivity not evaluated by most of the indicators used in health, It is therefore recommended to incorporate holistic and comprehensive care, incorporating individualized information about surgical options and freedom of choice and sexual education to the woman and her partner before surgery, to achieve an adequate quality of life.

Regarding the preparation of women who will undergo hysterectomy, the review of the literature reports barriers that include cultural and personal restrictions, the embarrassment of patients and physicians and low educational levels, which do not allow the clear delivery of information on definitions and consequences of surgery in the sexual sphere of women, addressing these problems without precision, both with the woman and with the sexual partner. Urrutia et al. reported different barriers perceived by hysterectomized women during the surgical process: technical language, lack of time, anger, contradictions in the indications and remoteness of health professionals; barriers in women: shyness, embarrassment, lack of confidence, fear and conformity; consequently, it is concluded that the challenge for health professionals is to develop appropriate communication techniques to improve health outcomes in this area.

It is so, that studies have recognized the relevance of providing patient education on the possible negative post-surgical effects in relation to sexual function, thus allowing acceptance of the surgical process and preventing complications. Along the same lines, researchers have reported the need for the person providing the information to be of the same sex, since this allows the woman to establish an adequate relationship between women and to have the freedom to ask questions.

However, few studies have been reported on the effect of nursing educational interventions aimed at hysterectomized women, although there is evidence that educational interventions can improve health-related behaviors, as reported by Hosseini et al. who, using the PRECEDE educational model (Predisposing, Reinforcing and Enabling Constructs in Educational Diagnosis and Evaluation), achieved a significant improvement in the experimental group about the control group in all the domains of sexual function. In addition to this, improvement has been evidenced through psychoeducational programs preventing emotional alterations and sexual dysfunctions, also favoring physical and emotional recovery, a return to a satisfactory active sexual life.

Research problem:

What is the significance of education in the perioperative period, in women undergoing hysterectomy? How efficient is a self-care-based nursing educational intervention for the improvement of health-related quality of life, sexual function, and self-esteem in women undergoing hysterectomy for a benign cause? 2 FRAME OF REFERENCE 1.2.1 THEORETICAL-CONCEPTUAL FRAMEWORK 1.2.1.1 HYSTERECTOMY Hysterectomy is one of the most common surgical procedures in women after cesarean section, and in 2004, around 600,000 such surgical interventions were performed in the United States. In addition, the literature reports that the rate of hysterectomy has varied between 6.1 and 8.6 per 1000 women of all ages.

Hysterectomy is a surgical procedure that consists of the removal of the body of the uterus, with or without the cervix and its adnexa. It is performed using various techniques that vary in the level of intervention and the access route, which can be abdominal, vaginal, or a combination of the two. Currently, there is a trend towards the more frequent use of less invasive surgical procedures such as laparoscopy, which is minimally invasive, and robotics, in search of the possibility of preserving the greatest amount of healthy organs and tissues, since hysterectomy is a complex, multidimensional experience.

The most common indications for hysterectomy are fibroids or leiomyomas, abnormal bleeding, endometriosis, uterine prolapse and others. At least 80% of these procedures are indicated for the treatment of benign pathology of the female genital tract, being a surgical intervention that has been downplayed because it is considered a routine intervention in health services, contributing to the increase of its frequency.

It is worth mentioning that the removal of the uterus has a great significance for women, both in the regulation of sexual and physiological functions, as well as a source of energy, vitality and maintenance of youth. Hysterectomy, by putting an end to the reproductive stage of the woman, affects her femininity and can cause alterations in self-esteem, in the relationship with her partner, conflict with the social environment, among others.

1.2.1.2 SEXUAL FUNCTION Sexual function is the activity proper to each sex, it is constituted as the result of an activation process between stimulus and response and begins to function at birth and depends on several factors, especially factors of the sociocultural environment, which will determine masculine and feminine behaviors and learning.

The development of sexual function is complex, being necessary to understand it through elements that allow its conceptualization, as is the case of the Theory of the variability of sex and sexual function. This theory explains the variation that the human being may have concerning sexual aspects, taking into account the existence of internal limits, minor and major limits, which leads to adequate functioning. Thus, sexual functioning will be within the normal range.

1.2.1.3 SELF-ESTEEM Self-esteem is an agent of self-protection against risk situations in health, social interaction and productivity. It allows personal development to be achieved through positive thoughts, being a fundamental element to have perspectives in life and psychological well-being.

Self-esteem is built throughout the life of the human being, it gathers thoughts, feelings, sensations and experiences lived throughout life, having its greatest development in childhood and adolescence. Self-esteem is also shaped by the image that the human being has of himself, the relationships with his environment, his values and objectives.

1.2.1.4 HEALTH-RELATED LIFE QUALITY Quality of life is a complex, multifactorial concept that refers to well-being or life satisfaction and the relationship with aspects of social, physical and psychological functioning, and it is the appropriate interaction of these elements that determines the quality of life of individuals.

The term life quality has been included since the 1950 in the area of medicine and later in psychology. From that time to the present, the concept has undergone several modifications. In 1982 Kaplan and Bush proposed the term Health-Related Life Quality to distinguish the broad concept of Life Quality from those aspects specifically relevant to health status and health care.

1.2.1.5 OREM'S SELF-CARE DEFICIT THEORY In 1969, Orem defined Self-care as an existing activity and behavior directed by people towards themselves, others or the environment, determining that the quantity and quality of care improve people's well-being. Orem's theory considers basic care as the center of assistance to human beings to improve their well-being; this theory gives nursing a leading role since it allows knowing, acting and helping people to meet their needs and demands for self-care, when this capacity is insufficient in people.

To understand the development of Orem's theory, three specific theories were articulated: self-care, self-care deficit and nursing systems.

1.2.1.6. PLISSIT MODEL

There are theories and models that can be nuanced with others to achieve a favorable effect in the interventions proposed to women awaiting surgical resolution (hysterectomy) and thus the incorporation of the PLISSIT Model has been considered. This conceptual model, which facilitates the treatment of sexual problems, was developed by Annon in 1976. PLISSIT is an acronym and each letter or pair of letters designates a suggested method for managing presenting sexual concerns. The four levels are presented below:

1. P-Permission: refers to the first level of intervention and usually becomes the nurse's responsibility as the initial contact with the patient within the health care team.
2. LI-Limited information: this is the second level of intervention and refers to information on normal sexual functioning or detailed aspects of surgery, anesthesia, medications, activity, complications, among others.
3. SS-Specific suggestion: refers to the necessary and specific orientation and information related to the problems detected about the recovery of their sexual functioning, which may be related to fear, fear, among others. These suggestions can be so about the referral to another more specialized level.
4. IT-Intensive therapy: this is the last stage of the PLISSIT model and is recommended for couples who have undergone the three levels of intervention and have not been successful; this stage involves mental health professionals and sex therapists to promote satisfactory sexual relations between the woman and her partner.

1.2.1.7. THEORY FOR DESIGNING INTERVENTIONS The theory-based approach to intervention relies on the propositions of the middle-range theory underlying the problem to develop interventions.

The application of the theory-based approach to designing interventions involves the following steps:

Step 1: Conceptualizing the problem, refers to the necessary understanding of the problem derived from a middle-range nursing theory, taking into account the need to know the nature of the problem, how it manifests itself, its severity, causal factors, and consequence concerning the population of interest.

Step 2: Determine the aspects of the problem that will be the object of intervention, this step refers to identifying the aspects of the problem that are susceptible to change and become the target of the intervention.

Step 3: Outline the necessary intervention strategies that target the aspects of the presenting problem identified as amenable to change, maintaining consistency between the nature of the problem aspect and the intervention strategy essential to the design of problem treatments in a direct, effective and efficient manner.

Step 4: Select the mode of delivery and dosage of the intervention through a carefully selected medium to be consistent with the nature of the intervention strategies, and to facilitate the delivery of the active ingredients of the intervention in an appropriate form.

Step 5: Specify intervention elements to conceptualize and guide their operationalization in an intervention manual. The description of the elements allows the integration of information on active ingredients, mode of administration, and dosage.

1.2.1.8. NURSING TECHNOLOGY The new healthcare reality, given by the challenges that arise such as longer life expectancy, increase in chronic diseases, the emergence of new social problems, globalization, generate the need to seek strategies that facilitate greater management capacity, organization, and healthcare situation. Nursing professionals cannot stay away from new information and communication technologies (ICT), since these are useful tools to complement face-to-face care, allowing them to adapt to people's needs and guaranteeing the achievement of the care provided by nursing professionals.

1.2.3 EMPIRICAL FRAMEWORK For the present study, it was searched for research on the impact of hysterectomy on the women who undergo it and on the effectiveness of interventions to improve the life quality-related health, sexual function and self-esteem in women undergoing hysterectomy. It is worth mentioning that most of the research found refers to the development of surgical techniques related to oncological processes, leaving in the background the educational interventions that have addressed the benefits of pre- and post-surgical interventions to prevent complications in hysterectomized women. Regarding the latter, it has been reported that more evidence is needed regarding the inclusion of theoretical support for the development of future studies in the field of interventions.

The following is a synthesis of findings from the studies retrieved. First of all, studies that report the impact of hysterectomy on the study variables will be presented:

The literature shows the existence of individual differences in coping with the removal of the uterus in a woman, which may cause alterations in the psychological, physical, social and sexual dimensions, as shown in a review study in which 61% of women were affected in the emotional component and the sexual dimension after surgery, also recognizing the importance of providing formal sex education to women and partners before the surgery, to prevent post-surgical alterations.

In addition to this, in Iran the relationship between hysterectomy and sexual function was evaluated in a retrospective cohort study of 44 women, the results showed changes in sexual function including: decreased sexual pleasure during orgasm, increased vaginal dryness, increased vaginal contraction, there is also the fear of restarting sexual intercourse, which may occur due to psychological problems resulting from the family and sexual environment.

As it is possible to observe, the literature reports possible impact on the sexual functions of women, given by the total removal of the uterus and would be related to the shortening of the vaginal vault, uterovaginal alterations, among others, may affect the sexual function, significantly affecting the life quality.

The following is a synthesis of findings from studies that report on the effectiveness of interventions to improve health-related life quality, sexual function, and self-esteem in women undergoing hysterectomy:

It is worth mentioning that this last study has served as a basis to guide aspects in the elaboration of the intervention of the present research, allowing the identification of the educational needs of hysterectomized women, to promote the recovery of their health, by recognizing the predisposing factors, the reinforcing factors such as the family, the health team and the factors of availability of resources and skills for the result of the intervention. It was also important as a basis for the calculation of the population, the number of sessions, the duration time.

1.3 HYPOTHESIS Conceptual hypothesis 1: Hysterectomized women in the experimental group improve female sexual function after the nursing educational intervention for those in the comparison group.

Working hypothesis:

Hysterectomized women in the experimental group have better scores on the desire subscale of female sexual function after the nursing educational intervention than those in the comparison group.

Hysterectomized women in the experimental group had better scores on the sexual function arousal subscale after the nursing education intervention than those in the comparison group.

Hysterectomized women in the experimental group have better scores on the lubrication subscale of female sexual function after the nursing education intervention than those in the comparison group.

Hysterectomized women in the experimental group have better scores on the orgasm subscale of female sexual function after the nursing education intervention compared to those in the comparison group.

The hysterectomized women in the experimental group had better scores on the subscale satisfaction of female sexual function after the nursing education intervention than those in the comparison group.

The hysterectomized women in the experimental group have better scores in the pain subscale of female sexual function after the nursing education intervention than those in the comparison group.

Conceptual hypothesis 2: Hysterectomized women in the experimental group have a better health-related quality of life after the nursing education intervention than those in the comparison group.

Working hypothesis:

Hysterectomized women in the experimental group scored better on the physical health component of health-related quality of life after the nursing educational intervention relative to those in the comparison group.

Hysterectomized women in the experimental group scored better on the mental health component of health-related quality of life after the nursing education intervention than those in the comparison group.

Conceptual hypothesis 3:

Hysterectomized women in the experimental group present a higher level of general self-esteem after the nursing educational intervention compared with those in the comparison group.

1.4 GENERAL OBJECTIVE To know the significance of education in the perioperative period in women undergoing hysterectomy for benign causes.

To determine the efficacy of a nursing education intervention based on self-care in improving female sexual function, health-related quality of life and self-esteem in women undergoing hysterectomy for benign causes.

SPECIFIC OBJECTIVES

Concerning the hysterectomized women participating in the study:

1. To identify the educational needs of women in the perioperative stage of hysterectomy.
2. To describe the biosociodemographic profile of the experimental group and the comparison group.
3. To determine the female sexual function of the experimental group and comparison group in a pre-and post-test measurement.
4. To establish the health-related life quality of the experimental group and comparison group in a pre-and post-test measurement.
5. To determine the self-esteem of the experimental group and comparison group in a pre-and post-test measurement.
6. To evaluate the efficacy of the nursing educational intervention directed to the experimental group versus the traditional approach in the comparison group in relation to:

Female sexual function Health-Related Life Quality Self-esteem 2. SUBJECTS AND METHODS 2.1 STUDY DESIGN The design will be sequential exploratory mixed, which is composed of an initial phase of qualitative data collection and analysis and a final phase where quantitative data are collected and analyzed. This mixed mixture makes it possible to determine clear stages, being necessary to analyze the data thoroughly from one stage to the other.

In addition to the above, from the point of view of intervention design, this would be a Phase II study. This phase includes the initial comparison with a control group, which may produce preliminary evidence that the intervention has the desired effects, a better understanding of the theoretical frameworks, information about appropriate control groups, a specific intervention manual, the most appropriate outcome measures, and considerations for a Phase III trial.

2.1.1 QUALITATIVE PHASE Design The present study constitutes qualitative research which corresponds to a systematic and subjective methodological approach used to describe life experiences and give them meaning. This type of research produces descriptive data, with people's own words, in verbal or written form, and observable behavior.

This research will have a descriptive approach since for this study it is not required to penetrate deeply into the data, therefore, it has a low level of interpretation, therefore, it will summarize the phenomenon.

Participants The participants in this research are all those women who are in the perioperative period of hysterectomy attending the Isidro Ayora Gynecological and Obstetric Hospital (HGOIA): a specialized, teaching, third level hospital located in the province of Pichincha, city of Quito, and is a reference for the entire national territory, with 210 beds for gynecological, obstetric and neonatology hospitalization and is an operative unit of the Ministry of Public Health.

Sample The sample is a part of the study population. According to Burns and Grove, this type of sampling is one of the most commonly used in qualitative nursing research. In this type of sampling, the researcher will consciously select the participants, who in his opinion are representative to be included in the study, thus achieving a purposive sampling by convenience, since the thesis candidate will select those women who are in the perioperative period of hysterectomy and are living this experience.

Location The interviews will be conducted in the procedure room of the gynecology hospitalization service of the Isidro Ayora Obstetric Gynecology and Gynecology Hospital, being this a pleasant place without noise that favors a pleasant dialogue with the patient, to achieve an adequate interview. If the woman cannot attend the interview in person, the interview will be conducted virtually (video or telephone).

Data Collection Technique.-Semi-structured interview:

The interviews will be conducted by the researcher in an individualized manner in person or virtually. For this purpose, an interview guide will be available, which will have questions grouped by themes or categories, based on the objectives of the study. According to Cisterna, it is the researcher who gives meaning to the results of his research, one of the basic elements to be taken into consideration is the elaboration and distinction of topics from which the information is collected and organized. For this purpose, a distinction must be made between categories, which denote a topic in itself, and subcategories, which detail this topic in micro aspects. These categories and subcategories can be aprioristic, i.e., constructed before the data collection process.

Procedures (recruitment and data collection) Prior to the start of the study, the corresponding permits will be requested from the Isidro Ayora Obstetric and Gynecological Hospital. Subsequently, the study will be submitted to the consideration of the Scientific Ethical Committee of the Faculty of Nursing of the Universidad de Concepción, the Scientific Ethical Committee of the Vice-Rectory of Research and Development of the Universidad de Concepción, the Ethics Sub-Committee of the Universidad Central del Ecuador and the Teaching and Research Committee of the Isidro Ayora Gynecological-Obstetric Hospital. Once the approvals have been obtained, we will proceed to access the information of the patients who are in the pre-surgical period. The women will be contacted by telephone, inviting them to participate in the present study and the interview. If they agree to participate, an appointment will be made and will be alternated with the medical consultation, taking advantage of the hospital visit and the interview. In the case where the woman cannot attend the face-to-face interview, it will be conducted virtually (video or telephone).

Data coding In this study, the researcher will transcribe the recorded interviews. Once the transcript is available, the information will be selected according to the previously cataloged categories, which will be assigned an abbreviation to be coded and subsequently analyzed.

Data analysis

The interviews will be analyzed by the student using the content analysis technique proposed by Bardin:

1. Pre-analysis
2. Exploitation of the material
3. Processing of results. 2.1.2 QUANTITATIVE PHASE This study is a quasi-experimental, non-equivalent control group design. This type of design is used when it is difficult to randomize the groups, either because of adverse conditions in the context or logistical difficulties.

It is necessary to mention that this type of design can be used when it is desired to verify the efficacy of interventions, as in the case of the present study.

Since this is a quasi-experimental study, it will comply with the following characteristics.

The experimental group, which corresponds to women on the waiting list for gynecological surgery, will be intentionally exposed to the nursing educational intervention, which corresponds to the independent variable, in order to observe the variation in the dependent variables (female sexual function, health-related life quality and self-esteem).

The efficacy of the nursing educational intervention with technological support (independent variable) on the dependent variables (female sexual function, health-related life quality and self-esteem) will be measured.

The following is the outline of the design with a non-equivalent control group.

According to what has been previously stated, the conformation of groups would be as follows:

Comparison group It will consist of women between 35 and 65 years of age who are on the waiting list for surgical treatment (hysterectomy) at the gynecology service of the HGOLEA and receive routine care, which consists of assessment and registration of vital signs, physical examination, clinical gynecological assessment, review of complementary tests and general indications. Patients do not receive detailed instructions about preoperative care and preparation, sex education, complications, or resumption of normal activities. Upon discharge from the hospital, an outpatient postoperative consultation is scheduled after 8 days and one month.

Experimental group It will be made up of women between 35 and 65 years of age who are on the waiting list for surgical treatment (hysterectomy) in the gynecology service of the HGOIA. Women seen at this facility receive care similar to that previously described for the HGOLEA. This group will additionally receive the educational intervention of face-to- face nursing with technological support.

2.4 TECHNOLOGY-SUPPORTED FACE-TO-FACE NURSING EDUCATION INTERVENTIONS There are prior considerations for the development of protocols that contain interventions and are pilot studies, therefore they consist of essential thinking actions interconnected to the whole research process, which includes a clear definition of the problem, for which change is sought, specifying the population that is most at risk, determining the reasons why the problem occurs and identifying the problems most likely to change being the outcomes of interest, further quantifying the magnitude of change if possible and identifying current practices or approaches to address the problem.

The first thought process that was carried out was the identification and definition of the problem since any intervention that can be designed is to improve, reduce or alter any problem with relevance to public health, the profession and the discipline of nursing and was reflected at the beginning of this study.

The next step was to justify the intervention to a specific problem of a small group of the population, but nevertheless be the result of a social and personal effort, therefore, should be considered to address.

The next step was to specify the population of the problem area that is susceptible to risk as a result of the problem posed.

The identification of available and relevant conceptual theoretical frameworks continued with the review of empirical evidence, which will inform how and why the intervention will have an impact for this population.

The identification of the triggering or contributing factors of the problem are modifiable through the proposed intervention.

Identification of possible outcomes or measures as an effect of the intervention, for example, altered female sexual function as evidence shows this to be a primary outcome as a consequence of hysterectomy. Quantifying the potential for improvement of the interventional problem (small, medium and large) or subjective improvements.

After the basis for the collection of the information described above, the objectives of the intervention will be drafted, its theoretical basis accompanied by a breakdown of the operational component so that there is coherence between the objectives, goals, activities and proposed results, carrying out in detail the sessions and all its components.

The remaining step in the design of interventions is the delineation of the expected outcomes of the intervention and the mechanisms underlying the effects of the intervention, which are then translated and transferred to the practice setting.

The following is a preliminary proposal, based on a review of the literature, of the phases of development and implementation of the Nursing Education Intervention and its operational elements.

Once the diagnostic operations were established, a proposal for nursing diagnoses based on self-care deficits was developed to determine the results to be achieved through the prescriptive operations, which will be used for the implementation of regulatory operations and subsequent evaluation through the control operations described below:

Importantly, health care professionals (nurses, gynecologists and sexologists) who have years of experience in caring for women with benign gynecological pathologies will be consulted. The invited professionals will be consultants on the content and applicability time of the face-to-face sessions. Among the professionals, an expert sexologist, a gynecologist dedicated to women's health and the Deputy Director of Nursing of the HGOIA were considered. In addition, support will be provided by eHealth experts and information technology (IT) developers, as well as designers and content specialists who will collaborate with the project team with extensive experience in the development of technological tools at the Central University of Ecuador.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria Be a woman between 35 and 65 years old, with a partner, on the waiting list for surgery scheduling (two weeks prior to surgery date assignment), with benign pathology, who knows how to read and write and has internet access.

Exclusion Criteria:

* Women with oncological pathology, complications or obstetric indication, with ectopic pregnancy, with oophorectomy, with mental illness or dementia, with a combination of several surgical procedures or some degree of physical or cognitive disability.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Female sexual function | 12 weeks and corresponds to the perioperative period for hysterectomy.
  The primary outcome expected from the intervention is the following to change Female Sexual Function in the hysterectomized woman. It will be measured with the Female Sexual Function Index, to achieve a score greater than 26 in the total sum of all domains, since a score less than 26 means sexual dysfunction.

SECONDARY OUTCOMES:
Health-related quality of life | 12 weeks and corresponds to the perioperative period for hysterectomy.
  Health-related quality of life. It will be measured with the Spanish version of the Health Questionnaire and the scores are from 0-100, and excellent is equal to 100.
Self-Steem | 12 weeks and corresponds to the perioperative period for hysterectomy.
  Self-Steem It will be measured with the Rosenberg Scale.The score is from 0 to 40, from 30 to 40 is high self-esteem, less than 25 low self-esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecological-Obstetric Hospital Isidro Ayora, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De La Cruz MS, Buchanan EM. Uterine Fibroids: Diagnosis and Treatment. Am Fam Physician. 2017 Jan 15;95(2):100-107. PMID 28084714
- [Result] Brill AI. Hysterectomy in the 21st century: different approaches, different challenges. Clin Obstet Gynecol. 2006 Dec;49(4):722-35. doi: 10.1097/01.grf.0000211946.51712.42. PMID 17082670
- [Result] Williams RD, Clark AJ. A qualitative study of women's hysterectomy experience. J Womens Health Gend Based Med. 2000;9 Suppl 2:S15-25. doi: 10.1089/152460900318731. PMID 10714742
- [Result] Hammer A, Rositch AF, Kahlert J, Gravitt PE, Blaakaer J, Sogaard M. Global epidemiology of hysterectomy: possible impact on gynecological cancer rates. Am J Obstet Gynecol. 2015 Jul;213(1):23-29. doi: 10.1016/j.ajog.2015.02.019. Epub 2015 Feb 25. PMID 25724402
- [Result] Prusty RK, Choithani C, Gupta SD. Predictors of hysterectomy among married women 15-49 years in India. Reprod Health. 2018 Jan 5;15(1):3. doi: 10.1186/s12978-017-0445-8. PMID 29304867
- [Result] Brolmann HA, Bijdevaate AJ, Vonk Noordegraaf A, Janssen PF, Huirne JA. Hysterectomy or a minimal invasive alternative? A systematic review on quality of life and satisfaction. Gynecol Surg. 2010 Sep;7(3):205-210. doi: 10.1007/s10397-010-0589-9. Epub 2010 May 22. PMID 20700519
- [Result] Dawood NS, Mahmood R, Haseeb N. Comparison of vaginal and abdominal hysterectomy: peri- and post-operative outcome. J Ayub Med Coll Abbottabad. 2009 Oct-Dec;21(4):116-20. PMID 21067042
- [Result] Danesh M, Hamzehgardeshi Z, Moosazadeh M, Shabani-Asrami F. The Effect of Hysterectomy on Women's Sexual Function: a Narrative Review. Med Arch. 2015 Dec;69(6):387-92. doi: 10.5455/medarh.2015.69.387-392. PMID 26843731
- [Result] Demirtas B, Pinar G. Determination of sexual problems of Turkish patients receiving gynecologic cancer treatment: a cross-sectional study. Asian Pac J Cancer Prev. 2014;15(16):6657-63. doi: 10.7314/apjcp.2014.15.16.6657. PMID 25169504
- [Result] Lonnee-Hoffmann R, Pinas I. Effects of Hysterectomy on Sexual Function. Curr Sex Health Rep. 2014;6(4):244-251. doi: 10.1007/s11930-014-0029-3. PMID 25999801
- [Result] Dukeshire S, Gilmour D, MacDonald N, MacKenzie K. Development and evaluation of a web site to improve recovery from hysterectomy. Comput Inform Nurs. 2012 Mar;30(3):164-75; quiz 176-7. doi: 10.1097/NCN.0b013e31823eb8f9. PMID 22266705
- [Result] Katz A. Sexuality after hysterectomy: a review of the literature and discussion of nurses' role. J Adv Nurs. 2003 May;42(3):297-303. doi: 10.1046/j.1365-2648.2003.02619.x. PMID 12680974
- [Result] Vonk Noordegraaf A, Huirne JA, Pittens CA, van Mechelen W, Broerse JE, Brolmann HA, Anema JR. eHealth program to empower patients in returning to normal activities and work after gynecological surgery: intervention mapping as a useful method for development. J Med Internet Res. 2012 Oct 19;14(5):e124. doi: 10.2196/jmir.1915. PMID 23086834
- [Result] Varsi C, Ekstedt M, Gammon D, Ruland CM. Using the Consolidated Framework for Implementation Research to Identify Barriers and Facilitators for the Implementation of an Internet-Based Patient-Provider Communication Service in Five Settings: A Qualitative Study. J Med Internet Res. 2015 Nov 18;17(11):e262. doi: 10.2196/jmir.5091. PMID 26582138
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Schmitt DP, Allik J. Simultaneous administration of the Rosenberg Self-Esteem Scale in 53 nations: exploring the universal and culture-specific features of global self-esteem. J Pers Soc Psychol. 2005 Oct;89(4):623-42. doi: 10.1037/0022-3514.89.4.623. PMID 16287423
- [Result] Ware JE Jr. Methodology in behavioral and psychosocial cancer research. Conceptualizing disease impact and treatment outcomes. Cancer. 1984 May 15;53(10 Suppl):2316-26. doi: 10.1002/cncr.1984.53.s10.2316. PMID 6367942
- [Result] Vitale AT, O'Connor PC. The effect of Reiki on pain and anxiety in women with abdominal hysterectomies: a quasi-experimental pilot study. Holist Nurs Pract. 2006 Nov-Dec;20(6):263-72; quiz 273-4. PMID 17099413
- [Result] Dixon KD, Dixon PN. The PLISSIT Model: care and management of patients' psychosexual needs following radical surgery. Lippincotts Case Manag. 2006 Mar-Apr;11(2):101-6. doi: 10.1097/00129234-200603000-00008. PMID 16582703
- [Result] Brandsborg B, Nikolajsen L. Chronic pain after hysterectomy. Curr Opin Anaesthesiol. 2018 Jun;31(3):268-273. doi: 10.1097/ACO.0000000000000586. PMID 29474214
- [Result] Goetsch MF. The effect of total hysterectomy on specific sexual sensations. Am J Obstet Gynecol. 2005 Jun;192(6):1922-7. doi: 10.1016/j.ajog.2005.02.065. PMID 15970852
- [Result] Berlit S, Tuschy B, Wuhrer A, Jurgens S, Buchweitz O, Kircher AT, Sutterlin M, Lis S, Hornemann A. Sexual functioning after total versus subtotal laparoscopic hysterectomy. Arch Gynecol Obstet. 2018 Aug;298(2):337-344. doi: 10.1007/s00404-018-4812-7. Epub 2018 Jun 14. PMID 29948170
- [Result] Brandsborg B, Dueholm M, Nikolajsen L, Kehlet H, Jensen TS. A prospective study of risk factors for pain persisting 4 months after hysterectomy. Clin J Pain. 2009 May;25(4):263-8. doi: 10.1097/AJP.0b013e31819655ca. PMID 19590472
- [Result] Cheung LH, Callaghan P, Chang AM. A controlled trial of psycho-educational interventions in preparing Chinese women for elective hysterectomy. Int J Nurs Stud. 2003 Feb;40(2):207-16. doi: 10.1016/s0020-7489(02)00080-9. PMID 12559144
- [Result] Devine EC. Effects of psychoeducational care for adult surgical patients: a meta-analysis of 191 studies. Patient Educ Couns. 1992 Apr;19(2):129-42. doi: 10.1016/0738-3991(92)90193-m. PMID 1299818
- [Result] Vonk Noordegraaf A, Anema JR, van Mechelen W, Knol DL, van Baal WM, van Kesteren PJ, Brolmann HA, Huirne JA. A personalised eHealth programme reduces the duration until return to work after gynaecological surgery: results of a multicentre randomised trial. BJOG. 2014 Aug;121(9):1127-35; discussion 1136. doi: 10.1111/1471-0528.12661. Epub 2014 Feb 11. PMID 24511914
- [Result] van der Meij E, Huirne JA, Bouwsma EV, van Dongen JM, Terwee CB, van de Ven PM, den Bakker CM, van der Meij S, van Baal WM, Leclercq WK, Geomini PM, Consten EC, Schraffordt Koops SE, van Kesteren PJ, Stockmann HB, Ten Cate AD, Davids PH, Scholten PC, van den Heuvel B, Schaafsma FG, Meijerink WJ, Bonjer HJ, Anema JR. Substitution of Usual Perioperative Care by eHealth to Enhance Postoperative Recovery in Patients Undergoing General Surgical or Gynecological Procedures: Study Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2016 Dec 21;5(4):e245. doi: 10.2196/resprot.6580. PMID 28003177
- [Result] van der Meij E, Anema JR, Leclercq WKG, Bongers MY, Consten ECJ, Schraffordt Koops SE, van de Ven PM, Terwee CB, van Dongen JM, Schaafsma FG, Meijerink WJHJ, Bonjer HJ, Huirne JAF. Personalised perioperative care by e-health after intermediate-grade abdominal surgery: a multicentre, single-blind, randomised, placebo-controlled trial. Lancet. 2018 Jul 7;392(10141):51-59. doi: 10.1016/S0140-6736(18)31113-9. Epub 2018 Jun 21. PMID 29937195
- [Result] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Result] Bernhard LA. Sexuality and sexual health care for women. Clin Obstet Gynecol. 2002 Dec;45(4):1089-98. doi: 10.1097/00003081-200212000-00017. No abstract available. PMID 12438887
- [Result] Duncan LE, Lewis C, Jenkins P, Pearson TA. Does hypertension and its pharmacotherapy affect the quality of sexual function in women? Am J Hypertens. 2000 Jun;13(6 Pt 1):640-7. doi: 10.1016/s0895-7061(99)00288-5. PMID 10912747
- [Result] Enzlin P, Mathieu C, Vanderschueren D, Demyttenaere K. Diabetes mellitus and female sexuality: a review of 25 years' research. Diabet Med. 1998 Oct;15(10):809-15. doi: 10.1002/(SICI)1096-9136(199810)15:103.0.CO;2-Z. PMID 9796879
- [Result] den Bakker CM, Schaafsma FG, van der Meij E, Meijerink WJ, van den Heuvel B, Baan AH, Davids PH, Scholten PC, van der Meij S, van Baal WM, van Dalsen AD, Lips DJ, van der Steeg JW, Leclercq WK, Geomini PM, Consten EC, Schraffordt Koops SE, de Castro SM, van Kesteren PJ, Cense HA, Stockmann HB, Ten Cate AD, Bonjer HJ, Huirne JA, Anema JR. Electronic Health Program to Empower Patients in Returning to Normal Activities After General Surgical and Gynecological Procedures: Intervention Mapping as a Useful Method for Further Development. J Med Internet Res. 2019 Feb 6;21(2):e9938. doi: 10.2196/jmir.9938. PMID 30724740
- [Result] Kim H, Sefcik JS, Bradway C. Characteristics of Qualitative Descriptive Studies: A Systematic Review. Res Nurs Health. 2017 Feb;40(1):23-42. doi: 10.1002/nur.21768. Epub 2016 Sep 30. PMID 27686751
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801